CLINICAL TRIAL: NCT06387537
Title: Effects of Scapular Mobilization on Shoulder Proprioception and Pain in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUI/CTR/2024/2
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Adhesive Capsulitis
Keywords: Chronic pain, proprioception, scapular mobilization
MeSH Terms: conditions — Bursitis; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive conventional physical therapy and the second will receive conventional physical therapy along with scapular mobilization. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Conventional Physical Therapy ) (Active Comparator): Patients in this group will receive conventional physical therapy including Hot pack for 10 to 15 minutes, ROM exercises such as Internal & external rotation, Extension in standing, Pulley for elevation in sitting or standing, Forward flexion in supine using own head, pendulum (1min clockwise, 1 min anti clock wise),these are Low intensity, short duration, 1-5 sec, 2-3 times/day, pain free passive, AAROM.
  GH mobilization: kaltenborn low grade mobilization (grade I or II) for (1 minute), Then mobilization with movement 3 sets of 10 reps with 1 minute rest in between will be given.Strengthening exercises include Isometric in all planes, 5 second holds, 1 set of 10 each direction, against wall. Every session will be given for 30 minutes and a total of 12 sessions would be conducted over a period of 4 weeks.
  Interventions: Procedure: Conventional physical therapy
- Group B (Conventional physical therapy and Scapular mobilization) (Experimental): Patients will receive scapular mobilization in addition to conventional physical therapy including Hot pack for 10 to 15 minutes , ROM exercises such as Internal & external rotation, Extension in standing, Pulley for elevation in sitting or standing, Forward flexion in supine using own head, pendulum (1min clockwise, 1 min anti clock wise),these are Low intensity, short duration, 1-5 sec, 2-3 times/day, pain free passive, AAROM. GH mobilization: kaltenborn low grade mobilization (grade I or II) for (1 minute), Then mobilization with movement 3 sets of 10 reps with 1 minute rest in between will be given. Strengthening exercises include Isometric in all planes, 5 second holds, 1 set of 10 each direction, against wall.
  Scapular Mobilizations Glides- superior, inferior, distraction, upward and downward rotation (5 sets, 10 reps, 30 sec break in 1 session).Every session will be given for 30 minutes and a total of 12 sessions would be conducted over a period of 4 consecutive weeks.
  Interventions: Procedure: Conventional physical therapy; Procedure: Scapular mobilization.

INTERVENTIONS:
Procedure: Conventional physical therapy — Patients in this group will recieve hot pack, ROM exercises, strengthening exercises and Kaltenborn mobilizations. A total of 12 sessions, 3 sessions per week for 4 consecutive weeks. Sets and repetitions will be increased progressively.
Procedure: Scapular mobilization. — Scapular Mobilizations: Glides- superior, inferior, distraction, upward and downward rotation (5 sets, 10 reps, 30 sec break in 1 session).Every session will be given for 30 minutes and a total of 12 sessions would be conducted over a period of 4 consecutive weeks.
  Arms: Group B (Conventional physical therapy and Scapular mobilization)

SUMMARY:
Adhesive capsulitis is a common musculoskeletal condition. Painful gradual loss of both active and passive gleno-humeral motion resulting from progressive fibrosis and ultimate contracture of the gleno-humeral joint capsule.Scapular position and movement perception both effected by shoulder adhesive capsulitis, change in the scapular kinematics in the form of an increase in scapular lateral rotation, and reduced joint sense for shoulder movements in adhesive capsulitis. Physiotherapists have a wide range of options in managing Adhesive capsulitis including Electrotherapeutic modalities, kaltenborn mobilization, Maitland's mobilization,Mulligan's mobilization and Manipulation. So far studies have shown the efficacy of different treatments in combination or in isolation.Few studies on proprioception in rotator cuff tear, sub acromial impingment syndrome, but no obseved effects of scapular mobilization on shoulder proprioception in patients with adhesive capsulitis.Physical therapist focus on lowering pain and ROM limitations in the shoulder,but often neglect to evaluate proprioception/joint position sense as well as the roleof scapula in adhesive capsulitis during treatment.If found effective,this study can help in probviding treatment protocols for improving proprioception in patients with adhesive capsulits.

DETAILED DESCRIPTION:
Adhesive capsulitis is a common MSK condition with an insidious onset accompanied by stiffness and trouble sleeping on the affected side.This condition effects General population 2-5% globally, diabetics 10-20%. Women have a significantly higher incidence males 70% of cases are female.Adhesive capsulitis is a painful, gradual loss of both active and passive gleno-humeral motion resulting from progressive fibrosis and ultimate contracture of the gleno-humeral joint capsule.

The deficit in shoulder proprioception associated to pain and destruction to specific tissues including labrum, peri-capsular m/s ligaments & joint capsule.Scapular position and movement perception both affected by shoulder adhesive capsulitis, change in the scapular kinematics in the form of an increase in scapular lateral rotation, and reduced joint sense for shoulder movements in adhesive capsulitis.

Scapulothoracic joint mobilization improve kinematic of shoulder including scapulohumeral rhythm. This mobilization changes the relative position of scapula and reduce stress on Gleno-humeral joint.There are still many unanswered questions in the domain of position and movement senses, particularly with regard to rehabilitation of shoulder proprioception in patients with adhesive capsulitis.

Hence the current study will investigate the effects of scapular mobilization on shoulder proprioception and pain in patients with adhesive capsulitis.

This study includes Subjects with nonspecific adhesive capsulitis without specific identifiable etiology (i.e. infection, inflammatory disease) ,40-65 years of age both males and females and chronic shoulder pain > 3 months.The selection of subjects will be using non-probability purposive sampling technique.Participants will be randomized using sealed envelope method and allocated to one of the 2 groups.

The data collection tools for pain is VAS, for ROM and PROPRIOCEPTION is Goniometer and for disability is SPADI.

The time duration for treatment protocol is total of 12 sessions, 3 sessions per week for 4 consecutive weeks for approximately 25-30 mins.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Nonspecific adhesive capsulitis without specific identifiable etiology (i.e. infection, inflammatory disease)
* 40-65 years of age both males and females.
* Chronic shoulder pain > 3 months.

Exclusion Criteria:

* Patients with other shoulder joint pathologies, such as fractures or dislocations, glenohumeral instability or rotator cuff pathologies in the affected shoulder.
* Subjects who have undergone surgery or have experienced an acute trauma to the shoulder.
* Individuals with current or history of neurological disorders (such as stroke, Alzheimer's, or Parkinson's), rheumatologic diseases (such as rheumatoid arthritis or systemic lupus erythematous), or systemic illnesses (such as thyroid disease).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder Proprioception | 4 weeks
  Proprioception will be measured using the universal Goniometer which is 0 to 180 degree for half circle model or 0 to 360 degree for full circle models.
Pain Intensity | 4 weeks
  Pain will be assessed using Visual Analog scale which is 0-100 item scale.

SECONDARY OUTCOMES:
Shoulder Range of motion | 4 weeks
  Range of motion will be assessed using universal goniometer.
Shoulder Disability | 4 weeks
  Shoulder Disability will be assessed using shoulder pain and disability index.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan